CLINICAL TRIAL: NCT02334631
Title: A Double Blind Randomized Controlled Trial of High Volume Simethicone to Improve Visualization During Capsule Endoscopy
Brief Title: High Volume Simethicone VCE Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Sai Lai Sey, MD, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 7339
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Small Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume simethicone (Experimental): High volume simethicone is defined as 1125 mg simethicone in 750 ml of water (1.5 mg/ml).
  Interventions: Drug: High Volume Simethicone
- Standard volume simethicone (Active Comparator): Standard volume simethicone is defined as 300 mg simethicone in 200 ml of water (1.5 mg/ml).
  Interventions: Drug: Standard Volume Simethicone

INTERVENTIONS:
Drug: High Volume Simethicone — High volume simethicone is defined as 1125 mg simethicone in 750 ml of water (1.5 mg/ml).
  Arms: High volume simethicone
Drug: Standard Volume Simethicone — Standard volume simethicone is defined as 300 mg simethicone in 200 ml of water (1.5 mg/ml).
  Arms: Standard volume simethicone

SUMMARY:
Video capsule endoscopy (VCE) is a procedure where a small camera is swallowed to examine the small bowel. Although the procedure is useful for diagnosing small bowel diseases, air bubbles can obscure the recorded images. Simethicone is a medication that can be used to disperse the air bubbles. However, prior studies using this medication have shown only a modest benefit. In our study, we would like to investigate whether increasing the amount of medication will improve the recorded images further.

DETAILED DESCRIPTION:
BACKGROUND:

While VCE has become an important diagnostic tool for clinical practice, optimal preparation for VCE has yet to be determined.(13) The European Society of Gastrointestinal Endoscopy recommends bowel preparation but does not provide further details.(2) The Canadian Association of Gastroenterology, American Society of Gastrointestinal Endoscopy, American College of Gastroenterology, and American Gastroenterological Association make no specific recommendation. Many studies have addressed this knowledge gap, testing various regimens of purgatives.(14-18) A meta-analysis found that polyethylene glycol provided adequate visual quality in 68% of patients compared to 48% with fasting alone, while diagnostic yield climbed from 36% to 46%.(4) In contrast, oral preparation for colonoscopy produces adequate visualization in greater than 90% of patients.(19)

Intraluminal debris, bile, and air bubbles impair the visibility of small bowel mucosa during VCE. Simethicone, an anti-foaming agent, has been used with mixed success to improve image quality. Three studies investigated the addition of simethicone (30 mg, 600 mg, and 800 mg) to overnight fast, PEG, or mannitol demonstrated improvement in visualization with high preparation scores favouring the addition of simethicone.(7-9) In contrast, Wei and colleagues (10) compared simethicone (300 mg) + PEG with PEG alone and found that although simethicone improved visualization, adequate visualization was achieved in only 63% of patients. Similarly, Ge et al. (11) compared simethicone (300 mg) against fasting alone and found improvement in visualization with simethicone but this was limited to the proximal half of the small bowel and adequate visualization was limited to 55% of cases. Lastly, Rosa et al. (12) compared simethicone (100 mg) + PEG with PEG alone and did not find a difference in visualization score.

A potential reason for inconsistent improvement in small bowel visualization may be due to an inadequate volume of simethicone being delivered into the small bowel, especially the distal portions. Prior volumes of simethicone were small (<200 ml) and may have pooled in the stomach and become diluted by gastric juices before being delivered into the duodenum. Our hypothesis is that high volume simethicone may overcome this problem and improve small bowel cleansing to facilitate improved visualization during VCE.

STUDY DESIGN:

This is a double blind randomized clinical trial evaluating high volume simethicone (750 ml at 1.5 mg/ml) versus standard volume simethicone (200 ml at 1.5 mg/ml) for CE. Randomization will be performed in blocks of varying sizes through a web based interface, Research Electronic Data Capture (REDCap), to ensure concealed allocation. Patients, physicians, and outcome assessors will be blinded to randomization allocation.

INTERVENTION:

All patients will take a standard small bowel preparation consisting of the following starting the day before the procedure: clear fluids starting at lunch, two liters of PEG at 8 PM, and fasting starting at midnight. Patients arrive in the endoscopy unit at 6:45 AM the following morning. Randomization is performed via REDCap and simethicone given as follows: those randomized to high volume simethicone will drink a 750 ml solution (1125 mg simethicone diluted in 750 ml of water, 1.5 mg/ml) and those randomized to standard volume simethicone will drink a 200 ml solution (300 mg simethicone diluted in 200 ml of water, 1.5 mg/ml) in identical non-transparent lidded cups sealed with tamper tape prepared by the hospital's Clinical Trials Pharmacy and administered to the patient by the research nurse. Regardless of randomization results, the solution will be consumed over a 5 minute period and the patient instructed to resume fasting for 30 minutes before swallowing the capsule. Adherence will be assessed by collection of the cups after ingestion.

After swallowing the capsule, the patient is discharged from the endoscopy unit, encouraged to remain active for the day, allowed to have clear fluids in 2 hours, a light meal in 4 hours, and to return the CE recorder to the endoscopy unit at 5 PM. Once the CE recorder is returned, the patient is discharged from the endoscopy unit and has completed the study. Subjects will be called by the study nurse 7 days later to assess for adverse events.

CE will be performed with the Given Imaging SB3 capsule and reviewed with the accompanying software, RAPID v8.3. Videos will be reviewed in a blinded fashion without knowledge of randomization results using the Park score.(41)

ELIGIBILITY:
Inclusion Criteria

1. Patients undergoing small bowel video capsule endoscopy

Exclusion Criteria

1. Patients with a contraindication to VCE (small bowel strictures, oropharyngeal dysphagia, pregnancy, patients who are not surgical candidates)
2. Endoscopic insertion of video capsule endoscope
3. Inpatient procedures for active GI bleeding
4. Patients with fluid restriction or who are unable to drink up to 900 ml of fluid within 10 minutes prior to the VCE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Visualization quality | Once during review of capsule images
  Visualization quality will be scored in a blinded fashion using a validated score developed by Park et al. (World J Gastroenterol 2010;16(7):875-80.) Representative images from the small bowel will be serially selected at five-minute intervals. Each image is evaluated for two parameters: the proportion of visualized mucosa (VM) and degree of obscuration (DO) by bubbles, debris etc. The proportion of visualized mucosa is scored on a three- point scale: > 75% = 3, 50% to 75% = 2, 25% to 50% = 1, <25% = 0. The degree of obscuration is also scored in a three point scale: < 5 % = 3, 5% to 25% = 2, 25% to 50% = 1, > 50 % = 0. Mean scores for each parameter are obtained by dividing the sum of all images scored by the number of images. Finally the average of the two parameters is calculated. Both the whole, proximal, and distal small bowel will be scored separately. The first half of the small bowel will be considered proximal while the second half will be considered distal.

SECONDARY OUTCOMES:
Visualized mucosa sub-score | Once during review of capsule images
  The 'Visualized Mucosa' sub-score of the visualization quality score described above.
Degree of obscuration sub-score | Once during review of capsule images
  The 'Degree of Obstruction' sub-score of the visualization quality score described above.
Diagnostic Yield | Once during review of capsule images
  A.The study will be considered 'diagnostic' if a clinically relevant lesion is found.
  B. The lesion may be clinically related to the referral indication or incidental.
  C. Lesions will be classified into: angioectasia, ulceration, stricture, polyp, mass, or other.
Study Completion Rate | Once during review of capsule images
  Study will be considered complete if the capsule passes into the cecum.
Gastric Emptying Time | Once during review of capsule images
  Defined as the time from the first gastric image until the first duodenal image.
Small Bowel Transit Time | Once during review of capsule images
  Defined as the time from the first duodenum image until the first cecal image
Adverse Events | Once 7 days after the procedure.
  Adverse events will be defined as new abdominal pain, diarrhea, constipation, bloating, and other between 0-7 days after the procedure that is different than pre-existing symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael SL Sey, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre- Victoria Campus, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sey M, Yan B, McDonald C, Segal D, Friedland J, Puka K, Jairath V. A randomized controlled trial of high volume simethicone to improve visualization during capsule endoscopy. PLoS One. 2021 Apr 1;16(4):e0249490. doi: 10.1371/journal.pone.0249490. eCollection 2021. PMID 33793636